CLINICAL TRIAL: NCT02721849
Title: Randomisierte Kontrollierte Studie Zur Wirkung Von Yoga Bei Chronischen Kopfschmerzen im Jugendalter
Brief Title: Yoga for Chronic Headache in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research Director, Universität Duisburg-Essen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 15-6736
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Tension Type Headache; Migraine
MeSH Terms: conditions — Tension-Type Headache; Migraine Disorders | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- adolescent yoga / parent control (Experimental): The adolescent will receive an 12 week yoga course, while one parent will only answer the questionnaires.
  Interventions: Behavioral: Yoga for adolescents
- adolescent waitlist / parent yoga (Experimental): One parent will participate in an 12 week yoga course, while the adolescent will receive the intervention after the follow-up period.
  Interventions: Behavioral: Yoga for parents
- adolescent yoga / parent yoga (Experimental): Both adolescent and parent will participate in an 12 week yoga course at the same time.
  Interventions: Behavioral: Yoga for adolescents; Behavioral: Yoga for parents
- adolescent waitlist / parent control (No Intervention): The adolescent will receive the intervention after the follow-up period, while one parent will only answer the questionnaires.

INTERVENTIONS:
Behavioral: Yoga for adolescents — 12 week hatha yoga course for adolescents
  Arms: adolescent yoga / parent control; adolescent yoga / parent yoga
Behavioral: Yoga for parents — 12 week hatha yoga course
  Arms: adolescent waitlist / parent yoga; adolescent yoga / parent yoga

SUMMARY:
A randomized controlled trial to investigate the efficacy of yoga on tension type headache and / or migraine in adolescents between 12 and 16 years, consisting of a four group design which includes an 12 week yoga course and a three-month follow-up period. Both adolescent and one parent will be randomized either to yoga or no treatment. Primary outcome will be pain frequency in adolescents considering pain catastrophizing of parents.

ELIGIBILITY:
Inclusion Criteria:

Adolescent:

* tension type headache and/or migraine minimum at 4 days per month
* willingness to participate at least 10 out of 12 yoga sessions
* physical and cognitive ability to participate in light physical, breathing and relaxation exercises
* good german language

Parents:

* willingness to participate at least 10 out of 12 yoga sessions
* physical and cognitive ability to participate in light physical, breathing and relaxation exercises
* good german language

Exclusion Criteria:

* pregnancy or lactation
* attending a yoga class within the last 3 months prior to the study

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pain frequency adolescent | Week 12
  Measurement of pain frequency after yoga intervention via headache diary

SECONDARY OUTCOMES:
Pain frequency adolescent | Week 24
  Measurement of pain frequency after follow-up period via headache diary
Pain duration adolescent | Week 12
  Measurement of pain duration after yoga intervention via headache diary
Pain duration adolescent | Week 24
  Measurement of pain duration after follow-up period via headache diary
Pain intensity adolescent | Week 12
  Measurement of pain intensity after yoga intervention via headache diary
Pain intensity adolescent | Week 24
  Measurement of pain intensity after follow-up period via headache diary
Quality of life adolescent self-assessment | Week 12
  Measurement of quality of life in self-assessment after yoga intervention via the kidscreen 27 questionnaire
Quality of life adolescent self-assessment | Week 24
  Measurement of quality of life in self-assessment after follow-up period via the kidscreen 27 questionnaire
Quality of life adolescent external assessment | Week 12
  Measurement of quality of life in external assessment by one parent after yoga intervention via the kidscreen 27 questionnaire
Quality of life adolescent external assessment | Week 24
  Measurement of quality of life in external assessment by one parent after follow-up period via the kidscreen 27 questionnaire
Pain disability adolescent self-assessment | Week 12
  Measurement of pain disability in self-assessment after yoga intervention via the paediatric pain disability index (P-PDI)
Pain disability adolescent self-assessment | Week 24
  Measurement of pain disability in self-assessment after follow-up period via the paediatric pain disability index (P-PDI)
Pain disability adolescent external assessment | Week 12
  Measurement of pain disability in external assessment by one parent after yoga intervention via the paediatric pain disability index (P-PDI)
Pain disability adolescent external assessment | Week 24
  Measurement of pain disability in external assessment by one parent after follow-up period via the paediatric pain disability index (P-PDI)
Pain coping adolescent | Week 12
  Measurement of pain coping in self-assessment after yoga intervention via the Paediatric Pain Coping Inventory Revise (PPCI-R)
Pain coping adolescent | Week 24
  Measurement of pain coping in self-assessment after follow-up period via the Paediatric Pain Coping Inventory Revise (PPCI-R)
Depression adolescent | Week 12
  Measurement of Depression in self-assessment after yoga intervention via the Depressions Inventar für Kinder und Jugendliche (DIKJ)
Depression adolescent | Week 24
  Measurement of Depression in self-assessment after follow-up period via the Depressions Inventar für Kinder und Jugendliche (DIKJ)
Stress adolescent | Week 12
  Measurement of Stress in self-assessment after yoga intervention via the Problem Questionnaire (PQ)
Stress adolescent | Week 24
  Measurement of Stress in self-assessment after follow-up period via the Problem Questionnaire (PQ)
Pain catastrophizing parents | Week 12
  Measurement of parents pain catastrophizing in self-assessment by one parent after follow-up period via the Pain Catastrophizing Scale for Parents (PCS-P)
Pain catastrophizing parents | Week 24
  Measurement of parents pain catastrophizing in self-assessment by one parent after follow-up period via the Pain Catastrophizing Scale for Parents (PCS-P)
Quality of life parents | Week 12
  Measurement of parents quality of life in self-assessment by one parent after yoga intervention via the WHO Quality of Life Bref questionnaire (WHOQol-Bref)
Quality of life parents | Week 24
  Measurement of parents quality of life in self-assessment by one parent after follow-up period via the WHO Quality of Life Bref questionnaire (WHOQol-Bref)
Depression parents | Week 12
  Measurement of parents depression in self-assessment by one parent after yoga intervention via the Beck-Depression-Inventar (BDI)
Depression parents | Week 24
  Measurement of parents depression in self-assessment by one parent after follow-up period via the Beck-Depression-Inventar (BDI)
Stress parents | Week 12
  Measurement of parents stress in self-assessment by one parent after yoga intervention via the Cohen's Perceived Stress Scale (PSS-10)
Stress parents | Week 24
  Measurement of parents stress in self-assessment by one parent after follow-up period via the Cohen's Perceived Stress Scale (PSS-10)
Adverse events adolescent | Week 12
  Adverse events within the yoga course period of adolescents
Adverse events parents | Week 12
  Adverse events within the yoga course period of parents

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Elisabeth Krankenhaus, Essen
  - Kinderkrankenhaus St. Marien, Landshut

IPD SHARING:
Plan to Share IPD: No